CLINICAL TRIAL: NCT04366908
Title: Prevention and Treatment With Calcifediol of COVID-19 Coronavirus-induced Acute Respiratory Syndrome (SARS)
Brief Title: Prevention and Treatment With Calcifediol of COVID-19 Induced Acute Respiratory Syndrome
Acronym: COVIDIOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Junta de Andalucia (Other Government); Dynamic Solutions (Industry); Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVIDIOL
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: SARS-CoV 2; COVID19; SARS (Severe Acute Respiratory Syndrome); Cytokine Release Syndrome; Cytokine Storm
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Cytokine Release Syndrome | interventions — glycine N-choloyltransferase; Calcifediol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - best available therapy (Active Comparator): The subject will be treated with the best available therapy, which will include any combination of drugs included in the current protocol of the Ministry of Health and/or complementary notes issued by the Spanish Agency of Medicines and Health Products (AEMPS).
  Interventions: Drug: BAT
- Treatment (Experimental): The subject will be treated with the best available therapy, which will include any combination of drugs included in the current protocol of the Ministry of Health and/or complementary notes issued by the Spanish Agency of Medicines and Health Products (AEMPS) plus Calcifediol caps. 266 µg. According to the pharmacokinetics of Calcifediol evaluated in an inflammatory model, the posology will be
  * Start: 2 capsules
  * Days 3, 7, 14, 21, 28: 1 capsule
  Interventions: Drug: BAT + Calcifediol

INTERVENTIONS:
Drug: BAT + Calcifediol — The subject will be treated with the best available therapy, which will include any combination of drugs included in the current protocol of the Ministry of Health and/or complementary notes issued by the Spanish Agency of Medicines and Health Products (AEMPS) plus Calcifediol caps. 266 µg. According to the pharmacokinetics of Calcifediol evaluated in an inflammatory model, the posology will be
  Start: 2 capsules Days 3, 7, 14, 21, 28: 1 capsule
  Arms: Treatment
Drug: BAT — The subject will be treated with the best available therapy, which will include any combination of drugs included in the current protocol of the Ministry of Health and/or complementary notes issued by the Spanish Agency of Medicines and Health Products (AEMPS).
  Arms: Control - best available therapy

SUMMARY:
The administration of Calcifediol in patients with COVID-19, will reduce the development of SARS and the worsening of the various phases of the syndrome. Reducing at least 25% in ICU admission and death from the process, reducing days of hospitalization, facilitating the recovery of the same, acting significantly and positively, in any of its phases throughout the natural history of illness.

As a treatment with extensive experience of clinical use, safe, inexpensive, and potentially very effective, it will have a highly efficient cost-benefit impact on the prevention of SARS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 90 years
* PCR confirmed diagnosis of COVID-19. As an alternative to PCR, a determination of antigens or any other test that in the future is considered equivalent to these in its diagnostic value may be accepted as evidence
* Radiological image compatible with inflammatory pleuropulmonary exudate or patients with onset of symptoms in the last 7 days and with an uncomplicated respiratory infection for outpatient follow-up.
* Signature of direct or delegated informed consent

Exclusion Criteria:

* Being treated with Calcifediol or Cholecalciferol in any of its presentations and dosages
* Intolerance or allergy to Calcifediol or its components
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Admission to Intensive Care Unit | At day 28.
  Proportion of subjects who enter the Intensive Care Unit
Death | At day 28.
  Proportion of subjects who die.

SECONDARY OUTCOMES:
Time from onset of symptoms to discharge of patients in conventional hospitalization | At day 28.
  Compare the time (in days) at discharge in newly hospitalized patients on non-invasive ventilation.
ICU - Time until admission | At day 28.
  In patients who, in the course of their evolution, required admission with mechanical ventilation in the ICU, time until admission to Intensive Care Unit
ICU - Time mechanical ventilation is removed | At day 28.
  In patients who, in the course of their evolution, required admission with mechanical ventilation in the ICU, time until mechanical ventilation is removed.
Evaluation of the inflammatory markers related with the disease | At day 28.
  Evaluation of the inflammatory markers related to IL disease. Blood samples will be collected and assessed in order to evaluate interleukins related with the interleukin storm using immunological tests.
Vitamin D metabolites | At day 28.
  Evaluation of the Vitamin D metabolites.
Evolution in SatO2 | At day 28.
  Compare the evolution in SatO2
Evolution in the Sat O2/FiO2 ratio. | At day 28.
  Compare the evolution in the Sat O2/FiO2 ratio
Evolution in the degree of dyspnea | At day 28.
  Compare the evolution in the degree of dyspnea using the analog Borg scale
Evolution of the improvement of radiological findings by simple radiology | At day 28.
  Compare the evolution of radiological findings by simple radiology in the recruited subjects since their beginning in the trial until they end the trial
Incidence of adverse events | At day 28.
  Incidence of adverse events related to medication and its administration.
Appearance of hemorrhagic or thrombotic phenomena | At day 28.
  Incidence in the appearance of hemorrhagic or thrombotic phenomena.

CONTACTS AND LOCATIONS:
Overall Officials: José López Miranda, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
All the information will be published and accessible. It will be also available on demand.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Since the end publication of the results.
Access Criteria: Contact uicec@imibic.org

REFERENCES:
- [Derived] Stroehlein JK, Wallqvist J, Iannizzi C, Mikolajewska A, Metzendorf MI, Benstoem C, Meybohm P, Becker M, Skoetz N, Stegemann M, Piechotta V. Vitamin D supplementation for the treatment of COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 24;5(5):CD015043. doi: 10.1002/14651858.CD015043. PMID 34029377